CLINICAL TRIAL: NCT02202486
Title: Investigation of the Blood-brain and Blood-dura Barrier Durin Migraine Attacks Using MRI
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Faisal Mohammad Amin, medical doctor, Glostrup University Hospital, Copenhagen
Other Study IDs: H-3-2012-073
Record Dates: First submitted 2014-07-17; First posted 2014-07-29 (Estimated); Last update posted 2014-07-29 (Estimated); Status verified 2014-07

CONDITIONS: Migraine With Aura; Migraine Without Aura; Chronic Migraine
MeSH Terms: conditions — Migraine with Aura; Migraine without Aura

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Creatinine, blood glucose, potassium, haemoglobin, erytrocyte profile
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Migraine with aura: Brain MRI
  Interventions: Other: Brain MRI
- Migraine without aura: Brain MRI
  Interventions: Other: Brain MRI
- Chronic migraine: Brain MRI
  Interventions: Other: Brain MRI

INTERVENTIONS:
Other: Brain MRI — Brain MRI with gadolinium contrast

SUMMARY:
Substudy 1 Blood-brain barrier breakdown has been proposed in migraine patients. Our hypothesis that we will test in this study is that the blood-brain barrier breaks down during migraine attacks but not out side attacks using MRI.

Substudy 2 Altered cerebral resting-state functional connectivity networks have been reported in migraine patients outside migraine attacks. What happens during migraine attacks has never been investigated. The hypothesis we will test is that pain related networks are affected during spontaneous attacks using functional MRI.

Substudy 3 Old studies report that cerebral blood flow (CBF) is altered in patients with migraine with aura, but not in those without aura. We hypothesize that CBF is altered regionally during attacks, which we will investigate in this study using arterial spin labeling (ASL).

Substudy 4 Structural changes using voxel-based morphometry (VBM) of the brain have been suggested but never investigated during migraine attacks. Our hypothesis is that pain related structures show altered VBM during spontaneous migraine attacks.

DETAILED DESCRIPTION:
Brain MRI during and outside migraine attacks.

Up to 600 patients will be recruited, who will be given a phone number that they can call when they get migraine attacks.

The study will continue until 20 patients with migraine with aura, 20 patients without aura, 20 patients with chronic migraine have completed the study.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of migraine with aura, migraine without aura, or chronic migraine according to the International Headache Society.
* written informed consent.
* use of anticonceptive method by women in childbearing age.

Exclusion Criteria:

* tension type headache more than 5/month during last year.
* tension type headache on the experimental day.
* use of antimigraine medication or pain-killer on the experimental day before MRI.
* pregnant or breastfeeding women.
* contraindications against MRI.
* history or clinical sign of cardio- or cerebrovascular disease.
* untreated severe mental disorder or drug abuse.
* other diseases or disorders interpreted, by the examining doctor, to interfere with participation in the study.
* not accepting information about potential accidental finding during experiment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Migraine patients.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2012-09; Primary Completion 2015-07 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Blood-brain barrier alteration during migraine attacks | Up to 1 year
Cerebral blood flow alteration during migraine attacks | Up to 1 year
Resting-state functional brain connectivity alteration during migraine attacks | Up to 1 year
Voxel-based morphometry alteration during migraine attacks | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Faisal M Amin, MD, Principal Investigator — Danish Headache Center, Glostrup Hospital
Locations (1):
- Danish Headache Center, Glostrup Hospital, Glostrup Municipality, Copenhagen, Denmark

REFERENCES:
- [Derived] Amin FM, De Icco R, Al-Karagholi MA, Raghava JM, Wolfram F, Larsson HBW, Ashina M. Investigation of cortical thickness and volume during spontaneous attacks of migraine without aura: a 3-Tesla MRI study. J Headache Pain. 2021 Aug 21;22(1):98. doi: 10.1186/s10194-021-01312-9. PMID 34418951